CLINICAL TRIAL: NCT03336346
Title: The Effect of Dolutegravir-based ART on Plasma Etonogestrel Levels in HIV-infected Women Using Contraceptive Implants in Botswana
Brief Title: Effect of Dolutegravir on Etonogestrel Levels in HIV-infected Women in Botswana
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor of Population and Family Health; Chief, Division of Family Planning & Preventive Services, Columbia University
Other Study IDs: AAAQ8556
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Contraceptive Usage; HIV Infections; Drug Interaction
Keywords: DTG; Dolutegravir; Efavirenz; Etonogestrel
MeSH Terms: conditions — Contraception Behavior; HIV Infections | interventions — dolutegravir; Electronystagmography; efavirenz

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- DTG group: Reproductive-aged HIV-infected women taking dolutegravir-based ART and using single-rod, etonogestrel-releasing, subdermal implant (ENG implant)
  Interventions: Drug: dolutegravir; Device: ENG implant
- No ART group: Reproductive-aged HIV-uninfected women using single-rod, etonogestrel-releasing, subdermal implant (ENG implant)
  Interventions: Device: ENG implant
- EFV group: Reproductive-aged HIV-infected women taking efavirenz-based ART and using single-rod, etonogestrel-releasing, subdermal implant (ENG implant)
  Interventions: Device: ENG implant; Drug: Efavirenz

INTERVENTIONS:
Drug: dolutegravir — HIV integrase strand transfer inhibitor used in combination ART
  Other Names: Tivicay; DTG
  Groups: DTG group
Device: ENG implant — Reversible contraception implant
  Other Names: Nexplanon ®; Implanon NXT ®; single-rod, etonogestrel-releasing, subdermal implant
Drug: Efavirenz — non-nucleoside reverse transcriptase inhibitor used in combination ART
  Other Names: Sustiva; EFV
  Groups: EFV group

SUMMARY:
The primary aim is to assess if etonogestrel (ENG) implant users taking dolutegravir (DTG) have a 20% or greater change in their ENG plasma levels, compared to women taking no antiretroviral therapy (ART). A secondary aim is to assess whether ENG implant users taking dolutegravir have significantly higher ENG plasma levels than ENG implant users taking efavirenz.

This is a cross-sectional, non-randomized evaluation to compare ENG levels between 3 and 12 months post-implant insertion in three groups of women: 1) women using DTG-based ART (n=90), 2) women using EFV-based ART (n=90), and 3) women using no ART (not HIV infected) (n=90). This study will be conducted in Botswana in Southern Africa among women using the ENG implant, and involves a one-time collection of blood and questionnaire.

DETAILED DESCRIPTION:
Efavirenz-based antiretroviral therapy is effective in treating HIV and had become standard in the World Health Organization (WHO) guidelines. However, despite its effectiveness in lowering viral load, there is also solid evidence that it decreases the effectiveness of etonogestrel-releasing implants. This presents a difficult clinical scenario in countries where the HIV burden is significant in reproductive age women.

Following the SINGLE trial, dolutegravir has replaced efavirenz in many settings as first-line ART. In 2016, Botswana became the first country in Africa to adopt this as a guideline, however, the effect that dolutegravir has on hormonal contraceptives has not been widely studied. This project seeks to understand the interaction between etonogestrel levels in HIV-infected women who are using dolutegravir-based ART by directly measuring etonogestrel blood levels using liquid chromatography-mass spectrometry in HIV-negative and HIV-infected women using contraceptive implants.

Because the implant is fairly new in Botswana, most participants will have had implants inserted 3-12 months prior to study. An HIV-infected, non-ART, comparison group is no longer permissible, practically or ethically, as countries across Africa, including Botswana, are moving to HIV "Test and Treat." This means that ART initiation is now occurring at time of HIV-diagnosis regardless of cluster of differentiation 4 (CD4) count or disease stage; therefore, in this study, the comparison group will be HIV-uninfected implant users. This comparison will answer the key question of whether the ENG implant when used simultaneously with DTG provides plasma ENG levels comparable to a group in which it has established contraceptive efficacy (i.e. HIV-uninfected, healthy women of reproductive age).

ELIGIBILITY:
Inclusion Criteria:

* Etonogestrel implant as their sole method of hormonal contraception
* Etonogestrel implant in-situ for three to twelve months.
* Dolutegravir (DTG) use for at least 60 days (Using DTG-based ART-regimen if applicable)
* Efavirenz (EFV) use for at least 60 days (Using EFV-based ART-regimen if applicable)

Exclusion Criteria:

* Exclude women using concomitant enzyme-inducing drugs, including rifampicin for tuberculosis treatment and anti-convulsant medications (phenytoin, carbamazepine, barbiturates, primidone, topiramate, oxcarbazepine)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive-aged HIV-infected women using dolutegravir and using single-rod, etonogestrel-releasing subdermal implant.
  Reproductive-aged HIV-infected women using efavirenz and using single-rod, etonogestrel-releasing subdermal implant.
  Reproductive-aged HIV-unifected women using single-rod, etonogestrel-releasing subdermal implant.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Difference (percentage) in ENG plasma levels in the DTG group compared to no ART group | Up to 12 months after implant
  Difference between the DTG group and no ART group

SECONDARY OUTCOMES:
Difference (percentage) in ENG plasma levels in the DTG group compared to EFV group | Up to 12 months after implant
  Difference between the DTG group and EFV group

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Westhoff, MD, Principal Investigator — Columbia University
Locations (1):
- Botswana-UPenn Partnership, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Undecided